CLINICAL TRIAL: NCT07007845
Title: The Effect of Osteopathy and Complete Vocal Technique on Phonation in Amateur Singers: A Crossover Study.
Brief Title: The Effect of Osteopathy and Complete Vocal Technique on Phonation in Amateur Singers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Complete Vocal Institute (Industry)
Collaborators: Buckinghamshire New University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CVT Support and Osteopathy
Record Dates: First submitted 2025-04-28; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Singing; Breathing Exercise; Osteopathy
Keywords: Diaphragm function; Singing technique; Support; Osteopathy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CVT Support optimisation (Active Comparator): The CVT Emergency Aid program focused on optimising the work on the diaphragm was conducted in 3 steps.
  Step 1 related to establishing diaphragmatic breathing by feeling expansion around lower ribs at inhalation.
  Step 2 related to establishing connection between pulmonary pressure and subtotal pressurisation by invoking inwards abdominal movements on controlled exhaled voiceless exercises (ssss-sound) Step 3 related to establishing dynamic control of subglottal pressure by performing fricative voice sounds (vvvf- and zzz-sounds) while contracting the abdominal wall inwards and thereby pressurising the pulmonary space leading to increased subglottal pressure on accents and extended pitch accents.
  Interventions: Behavioral: CVT Support intervention
- Osteopathy (Experimental): Osteopathic treatment: Dooming Diaphragm. The inferior costal margin was contacted with the hands, allowing the thumbs to rest just below the ribcage anteriorly. Care was taken to avoid contact with the xiphoid process, as this could cause discomfort for the patient. The patient was instructed to breathe deeply, and as they exhaled, gentle pressure was applied superiorly and laterally with the thumbs, rolling them underneath the ribcage as far as was comfortable. This process was repeated for 3-5 breath cycles or until no tension was felt in the thumbs during exhalation.
  Interventions: Procedure: Dooming Diaphragm

INTERVENTIONS:
Behavioral: CVT Support intervention — The CVT Emergency Aid program focused on optimising the work on the diaphragm was conducted in 3 steps. Step 1 related to establishing diaphragmatic breathing by feeling expansion around lower ribs at inhalation. Step 2 related to establishing connection between pulmonary pressure and subtotal pressurisation by invoking inwards abdominal movements on controlled exhaled voiceless exercises (ssss-sound) Step 3 related to establishing dynamic control of subglottal pressure by performing fricative voice sounds (vvvf- and zzz-sounds) while contracting the abdominal wall inwards and thereby pressurising the pulmonary space leading to increased subglottal pressure on accents and extended pitch accents.
  Other Names: CVT Support
  Arms: CVT Support optimisation
Procedure: Dooming Diaphragm — Osteopathic treatment: Dooming Diaphragm. The inferior costal margin was contacted with the hands, allowing the thumbs to rest just below the ribcage anteriorly. Care was taken to avoid contact with the xiphoid process, as this could cause discomfort for the patient. The patient was instructed to breathe deeply, and as they exhaled, gentle pressure was applied superiorly and laterally with the thumbs, rolling them underneath the ribcage as far as was comfortable. This process was repeated for 3-5 breath cycles or until no tension was felt in the thumbs during exhalation.
  Other Names: Osteopathic treatment of diaphragm
  Arms: Osteopathy

SUMMARY:
This study is about breathing function during singing, specifically aimed at improving the functionof the muscles in the respiratory system involved in control over the voice.The goal of the study is to examine if osteopathic techniques and/or work with support developedby Complete Vocal Institute influences voice quality and sense of ease using voice.The study compares two types of interventions:1: An osteopathic optimization treatment for diaphragm, a major muscle responsible for breathing.And2: A singing technique for learning stamina.Both techniques work on improving patterns of breathing which should make singing feel easier and lower future risks of injury and strain. The study takes place at Complete Vocal Institute where participant voices will be recorded by a microphone and by a laryngograph. In using the laryngograph, two gold-plated electrodes will be placed over the larynx. A microphone records the voice whereas EGG-electrodes record how the vocal folds are vibrating. Measurements are made before each type of treatment and after each treatment. Both are non-invasive and carry no risk to the voice. The recordings will be done in a sound-treated room for privacy.The singing intervention will involve breathing exercises, and the osteopathic treatment will involve a single fascia treatment. It is possible that the osteopathic treatment can leave participant diaphragms and the area around the lower ribs sore, this is normal and is expected to last no more than 24-48 hours. Each session is expected to last approximately one hour, and only a single visit will be required.To ensure comfort, please wear loose-fitting clothing that allows for easy breathing and singing. For one part of the intervention, participants will be asked to remove clothing like one would for any physical massage, so the therapist can access and treat the diaphragm.There are no costs involved nor compensation for participation in the study. Participation is completely voluntary. Should participants at any time wish to withdraw from the study, they are free to do so by informing Julie Bie at julie@netfyssen.dk hereof.All data will be anonymized and any information that could identify participants as a subject will be kept strictly confidential. No personal information will be included in the study report or other publication arising from the project analysis.If there have any questions, please contact the investigators at julie@netfyssen.dk or mathias@shout.dk. This research is being overseen by an Institutional Review Board ("IRB"). The two therapists involved in this study are insured, and the study has received favorable approval from the Ethics Committee of Buckinghamshire New University.

ELIGIBILITY:
Inclusion Criteria:

* General health, no known vocal pathology or ongoing respiratory infection
* No ongoing reflux symptoms
* Amateur singer

Exclusion Criteria:

* No prior osteopathic treatment related to voice
* No prior CVT Support Training

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2025-03-03 (Actual); Primary Completion 2025-03-07 (Actual); Study Completion 2025-04-28 (Actual)

PRIMARY OUTCOMES:
Maximum Phonation Time | Baseline
  The total amount in seconds a sustained phonation can be maintained
Mean sound pressure level | Baseline
  Sound pressure level, SPL, to indicate vocal loudness.
Maximum and minimum fundamental frequency | Baseline
  The maximum and minimum fundamental frequency as an indicator of singing note pitch.
Fx SD | Baseline
  Fundamental Frequency Standard Deviation (Fx SD)
Qx | Baseline
  Average Contact Quotient (Qx)
Jitter | Baseline
  Amount (in %) of Jitter during cycle to cycle variation of vocal fold oscillations on a sustained vowel measured by electroglottography
Normalised Noise Energy | Baseline
  Normalised Noise Energy (NNE) of acoustic radiated output during phonation
Cepstral Peak Prominence | Baseline
  Cepstral Peak Prominence (CPP) of sustained phonation
Maximum Phonation Time | Day 1
  The total amount in seconds a sustained phonation can be maintained
Mean sound pressure level | Day 1
  Sound pressure level, SPL, to indicate vocal loudness.
Maximum and minimum fundamental frequency | Day 1
  The maximum and minimum fundamental frequency as an indicator of singing note pitch.
Fx SD | Day 1
  Fundamental Frequency Standard Deviation (Fx SD)
Qx | Day 1
  Average Contact Quotient (Qx)
Jitter | Day 1
  Amount (in %) of Jitter during cycle to cycle variation of vocal fold oscillations on a sustained vowel measured by electroglottography
Normalised Noise Energy | Day 1
  Normalised Noise Energy (NNE) of acoustic radiated output during phonation
Cepstral Peak Prominence | Day 1
  Cepstral Peak Prominence (CPP) of sustained phonation
Maximum Phonation Time - post intervention | Day 1
  The total amount in seconds a sustained phonation can be maintained
Mean sound pressure level - post intervention | Day 1
  Sound pressure level, SPL, to indicate vocal loudness.
Maximum and minimum fundamental frequency - post intervention | Day 1
  The maximum and minimum fundamental frequency as an indicator of singing note pitch.
Fx SD - post intervention | Day 1
  Fundamental Frequency Standard Deviation (Fx SD)
Qx - post intervention | Day 1
  Average Contact Quotient (Qx)
Jitter - post intervention | Day 1
  Amount (in %) of Jitter during cycle to cycle variation of vocal fold oscillations on a sustained vowel measured by electroglottography
Normalised Noise Energy - post intervention | Day 1
  Normalised Noise Energy (NNE) of acoustic radiated output during phonation
Cepstral Peak Prominence - post intervention | Day 1
  Cepstral Peak Prominence (CPP) of sustained phonation

CONTACTS AND LOCATIONS:
Locations (1):
- Complete Vocal Institute, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
To respect the anonymity of study participants, data will not be shared beyond reasonable request that ensures privacy and GDPR compliance.